CLINICAL TRIAL: NCT04047823
Title: Relationships Between the Changes of Skin Temperature and Radiation Skin Injury
Brief Title: Temperature and Injury in Radiotherapy Radiation Skin Injury
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Han Xi Zhao, M.D.Ph.D, Shandong Cancer Hospital and Institute
Other Study IDs: FIR-2015
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Breast Neoplasm Female; Radiation Toxicity
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: a digital Infrared thermography (FLIR E5 Serial No.63985976） — Measurements were taken during radiation and additionally two weeks after radiotherapy weekly. Temperature change was measured by thermal infrared imager (FLIR) for 4 test areas within the supraclavicular radiation field and on an opposite non-irradiated area, which was outlined using a specific software package (FLIR Systems 6.3.17227.1001).

SUMMARY:
the main purpose of the present study was threefold: (1) to describe the thermographic response after radiation; (2) to investigate whether there was a significant temperature change over time and among the different radiation-dermatitis score; and (3) to test if temperature change could be used to predict the development of radiation-induced skin injury in the incipient stage.

DETAILED DESCRIPTION:
Radiation skin injury (RSI) is a frequent adverse reaction reported encountered by patients undergoing radiotherapy, occurring in about 87%-95% of irradiated patients and is characterized by swelling, redness, pigmentation, ulceration, fibrosis, pain, warmth, burning and itching of the skin. RSI has an effect on the level of discomfort experienced and the quality of life of patients, and may require interfering with radiation schedule and complex surgical reconstruction especially when combined with molecular targeted therapy. However, evaluation of RSI is not straightforward. There is no standard instrument for objective clinical evaluation of the severity of radiation skin injury.

Previous studies have shown that radiation leads to the development of cutaneous vasculature and generation of an inflammatory response, which will increased skin temperature. The skin temperature change due to laser or thermal injury has been measured in many studies with temperature and time as predictors of skin damage.

The most frequent method of skin temperature measurement has been the Infrared thermography. Consequently, the changes in the difference of skin temperature (DST) may be used as an objective, quantitative, and functional surrogate measure to determine and predict RSI.

ELIGIBILITY:
Inclusion Criteria:

* a pathologically proven breast cancer receiving three dimensional conformal radiated therapy followed by modified radical mastectomy
* ECOG PS≤1
* normal organ function
* no prior radiotherapy
* no concurrent chemotherapy

Exclusion Criteria:

* rash or unhealed wound in the radiation field,
* pregnancy or lactation
* the presence of connective tissue disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with a pathologically proven breast cancer receiving three dimensional conformal radiated therapy followed by modified radical mastectomy were eligible for the study. Other inclusion criteria included: age ≥18 years, ECOG PS≤1, normal organ function, no prior radiotherapy, and no concurrent chemotherapy.
  Exclusion criteria were as follows: rash or unhealed wound in the radiation field, pregnancy or lactation, and the presence of connective tissue disorder. All the enrolled were giving informed consent.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-10-02 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Thermographic response after radiation | during the radiotherapy
  Thermographic change were tested during radiation weekly
temperature changes among the different radiation-dermatitis score | during the radiotherapy
  temperature changes among the different radiation-dermatitis score acoording to RTOG score
temperature changes could be used to predict the development of dermatits in the incipient stage | during the radiotherapy
  Multiple linear regression analysis was performed to study the influence of various facters on severe dermatits.